CLINICAL TRIAL: NCT05052814
Title: Comparative Evaluation of the Effect of Three Different Root-canal Medicaments on Post-operative Pain in Re-treatment Cases: a Randomized Clinical Trial
Brief Title: The Effect of Root-canal Medicaments on Post-operative Pain in Re-treatment Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Hicran Dönmez Özkan, assistant professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/079
Record Dates: First submitted 2021-09-08; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Endodontically Treated Teeth
Keywords: retreatment
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calcium hydroxide ( Ca(OH)2 ) (Experimental): Root canal medicament which was placed into root canals with a lentulo spiral.
  Interventions: Other: root canal medicament-calcium hydroxide
- Chlorhexidine gel (CHX gel) (Experimental): Root canal medicament which was placed into root canals with a lentulo spiral.
  Interventions: Other: root canal medicament-chlorhexidine gel
- Calcium hydroxide+ CHX gel (Experimental): Root canal medicament which was placed into root canals with a lentulo spiral.
  Interventions: Other: root canal medicament-calcuim hyroxide &chlorhexidine ge

INTERVENTIONS:
Other: root canal medicament-calcium hydroxide — Two different root canal medicaments and their combination were placed into the root canals following the removal of previous root canal fillings and re-instrumentation. Afterward, postoperative pain scores were recorded at 6 and 12 hours and at 1, 2, 3, 4, 5, 6, and 7 days using the visual analog scale (VAS). Sensitivity on percussion, spontaneous pain, swelling, and antibiotic and analgesic requirements of the patients were married during clinical examinations performed postoperatively after 2 and 7 days.
  Arms: Calcium hydroxide ( Ca(OH)2 )
Other: root canal medicament-chlorhexidine gel — Two different root canal medicaments and their combination were placed into the root canals following the removal of previous root canal fillings and re-instrumentation. Afterward, postoperative pain scores were recorded at 6 and 12 hours and at 1, 2, 3, 4, 5, 6, and 7 days using the visual analog scale (VAS). Sensitivity on percussion, spontaneous pain, swelling, and antibiotic and analgesic requirements of the patients were married during clinical examinations performed postoperatively after 2 and 7 days.
  Arms: Chlorhexidine gel (CHX gel)
Other: root canal medicament-calcuim hyroxide &chlorhexidine ge — Two different root canal medicaments and their combination were placed into the root canals following the removal of previous root canal fillings and re-instrumentation. Afterward, postoperative pain scores were recorded at 6 and 12 hours and at 1, 2, 3, 4, 5, 6, and 7 days using the visual analog scale (VAS). Sensitivity on percussion, spontaneous pain, swelling, and antibiotic and analgesic requirements of the patients were married during clinical examinations performed postoperatively after 2 and 7 days.
  Arms: Calcium hydroxide+ CHX gel

SUMMARY:
This randomized clinical trial compares the effects of intracanal medicaments on the incidence of postoperative pain and flare-up in asymptomatic retreatment cases.

DETAILED DESCRIPTION:
Introduction: The aim of this study was to compare the effects of intracanal medicaments on the incidence of postoperative pain and flare-up in asymptomatic retreatment cases.

Methods: One hundred twenty patients with asymptomatic teeth with single-root, single-canal without spontaneous pain or swelling were included in the present study. All patients were previously undergone endodontic treatment but still had periapical radiolucencies. Patients were randomly and equally divided into three groups in which stratified randomization was performed based on the gender and the age of the patients. Intracanal medicaments were placed into the root canals following the removal of previous root canal fillings and re-instrumentation. Calcium hydroxide (Ca(OH)2), chlorhexidine gel (CHX), calcium hydroxide, and chlorhexidine gel combinations were used as intracanal medicaments in the present study. Postoperative pain scores were recorded at 6 and 12 hours and at 1, 2, 3, 4, 5, 6, and 7 days using a visual analog scale (VAS). Sensitivity on percussion, spontaneous pain, swelling, and antibiotic and analgesic requirements of the patients were evaluated during clinical examinations performed postoperatively after 2 and 7 days.

p.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 20 - 65 years of ages
2. Patients who agree to participate this study
3. Not taking analgesic or antibiotics in the last week
4. Single root and single-canal incisor, canine, premolar teeth that have been treated only once before
5. Teeth with previous endodontic treatment but with insufficient root canal filling on radiographic examination
6. Teeth with periapical lesions and at least 2 years since the previous treatment, although root canal filling seems sufficient
7. Periapical radiolucency, teeth with increased or unchanged according to pre-treatment radiography (if available)
8. Teeth are asymptomatic
9. Patients who had good oral hygiene

Exclusion Criteria:

1. Pregnant patients and patients in lactation period
2. Having used corticosteroids in the last 6 months
3. Individuals with systemic diseases (endocarditis, immune system diseases,etc.) requiring antibiotic prophylaxis
4. Having received immunosuppressive therapy within the last week
5. Patients who had systemic or allergic sensitivty for the NSAIDs and local ananesthetics
6. The presence of advanced periodontal disease (probing depth > 4 mm)
7. The presence of a foreign body in the root canal that prevents entry (broken file, post, etc.)
8. Fracture or crack in the root
9. Teeth that cannot reach the working length due to calcification in the root canal and step formation
10. Teeth that cannot be restored due to excessive loss of material in the coronal structure
11. The presence of more than one adjacent tooth requiring endodontic treatment that may cause reflected pain in the same patient.
12. Teeth that develop any complications ( breakage of endodontic file, perforation, inability to determine the working length with the apex finder) during the removal of the canal filling material.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-08-23 (Actual)

PRIMARY OUTCOMES:
Pain level comparison after the application of three different root canal medicaments in root canal : VAS (Visual Analogue Scale) at 6th hours. | 6 th hours
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after the application of three different root canal medicaments in root canal : VAS (Visual Analogue Scale) at 12 th hours. | 12 th hour
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after the application of three different root canal medicaments in root canal : VAS (Visual Analogue Scale) at 24th hours. | 24 th hour
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after the application of three different root canal medicaments in root canal : VAS (Visual Analogue Scale) at 2nd days. | 2nd days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after the application of three different root canal medicaments in root canal : VAS (Visual Analogue Scale) at 3th days. | 3th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after the application of three different root canal medicaments in root canal : VAS (Visual Analogue Scale) at 4th days. | 4th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after the application of three different root canal medicaments in root canal : VAS (Visual Analogue Scale) at 5th days. | 5th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after the application of three different root canal medicaments in root canal : VAS (Visual Analogue Scale) at 6th days. | 6th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.
Pain level comparison after the application of three different root canal medicaments in root canal : VAS (Visual Analogue Scale) at 7th days. | 7th days
  Based on the VAS (Visual Analogue Scale), the pain levels of the patients were assessed. The scale consisted of a 100-mm-long line divided into 10 equal intervals from 0 (no pain) to 100 (very severe pain). Every patient was asked to mark his or her perceived postoperative pain level on the line.

CONTACTS AND LOCATIONS:
Locations (1):
- Hicran Dönmez Özkan, Merkez, Aydın, Turkey (Türkiye)

REFERENCES:
- [Background] Erdem Hepsenoglu Y, Eyuboglu TF, Ozcan M. Postoperative Pain Intensity after Single- versus Two-visit Nonsurgical Endodontic Retreatment: A Randomized Clinical Trial. J Endod. 2018 Sep;44(9):1339-1346. doi: 10.1016/j.joen.2018.05.017. Epub 2018 Jul 24. PMID 30054099
- [Background] Gondim E Jr, Setzer FC, Dos Carmo CB, Kim S. Postoperative pain after the application of two different irrigation devices in a prospective randomized clinical trial. J Endod. 2010 Aug;36(8):1295-301. doi: 10.1016/j.joen.2010.04.012. Epub 2010 Jun 19. PMID 20647083